CLINICAL TRIAL: NCT02623166
Title: To Operationalise the Policy of Treating Uncomplicated Pneumonia, Diarrhoea and Fever in Children Aged 2-59 Months by Community Health Workers(CHW)
Brief Title: Treatment of Pneumonia, Diarrhoea and Fever in Children by Community Health Workers
Status: Completed | Type: Observational
Sponsor: Society for Applied Studies (Other)
Collaborators: World Health Organization (Other)
Responsible Party: Sponsor
Other Study IDs: 2015/517094-0
Record Dates: First submitted 2015-11-24; First posted 2015-12-07 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Pneumonia, Diarrhea, Fever
Keywords: Pneumonia; Fever; Diarrhoea
MeSH Terms: conditions — Pneumonia; Diarrhea; Fever

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators propose to test the feasibility and acceptability of community health workers (ASHAs and ANMs) being able to treat sick children in the community. There is a national policy for treatment for children aged 2-59 months with illnesses such as pneumonia, diarrhea and fever by community health workers (CHWs), this policy has not been implemented as yet in Haryana. This research will identify barriers and opportunities for use of CHWs as treatment sources.

DETAILED DESCRIPTION:
Using indepth interviews, focus group discussions and other qualitative research methods barriers and opportunities for promoting use of ASHAs as a treatment source for diarrhea, pneumonia and fever will be identified. An intervention package which includes training of ASHAs and ANMs to treat uncomplicated cases of pneumonia, diarrhea and fever, ensuring they have required supplies, creating awareness in community and monitoring and supervising the treatment provided by them will be implemented in primary health centre areas in Haryana, India. ASHAs will treat cases of fast breathing pneumonia with amoxicillin and refer children with danger signs or chest indrawing pneumonia. Three rounds of cross sectional surveys will be conducted to ascertain prevalence of morbidity, careseeking and hospitalizations in children aged 2 to 59 months.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2-59 months with uncomplicated pneumonia or diarrhoea or fever

Exclusion Criteria:

* Refusal for participation
* Diarrhea with dehydration
* Danger signs
* Chest indrawing pneumonia

Ages: 2 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study will be conducted in 2 primary health centres. These include 6 sub centres in Rasoolpur PHC (population ~57000) and 7 sub centres in Mandkola PHC (population ~57000).
Sampling Method: Non-Probability Sample
Enrollment: 24000 (Actual)
Dates: Start 2015-11; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Increase in the proportion of caregivers seeking care for 2-59 months old children with pneumonia, diarrhoea and fever from trained Community Health Workers (CHW) | To be assessed at baseline
Increase in the proportion of caregivers seeking care for 2-59 months old children with pneumonia, diarrhoea and fever from trained Community Health Workers (CHW) | To be assessed 5 months after start of study
Increase in the proportion of caregivers seeking care for 2-59 months old children with pneumonia, diarrhoea and fever from trained Community Health Workers (CHW) | To be assessed 8 months after start of study
Increase in proportion of caregivers seeking care for 2-59 months, old children with pneumonia, diarrhoea and fever from appropriate sources of care. | To be assessed at baseline
Increase in proportion of caregivers seeking care for 2-59 months, old children with pneumonia, diarrhoea and fever from appropriate sources of care. | To be assessed 5 months after start of study
Increase in proportion of caregivers seeking care for 2-59 months, old children with pneumonia, diarrhoea and fever from appropriate sources of care. | To be assessed 8 months after start of study

SECONDARY OUTCOMES:
Knowledge and perceptions of caregivers about treatment from trained CHWs assessed by indepth interviews and focus group discussions | To be assessed at baseline
Knowledge and perceptions of caregivers about treatment from trained CHWs assessed by indepth interviews and focus group discussions | To be assessed 5 months after start of study
Knowledge and perceptions of caregivers about treatment from trained CHWs assessed by indepth interviews and focus group discussions | To be assessed 8 months after start of study
Experiences of CHW about themselves as treatment providers assessed by indepth interviews using questionnaires | To be assessed at baseline
Experiences of CHW about themselves as treatment providers assessed by indepth interviews using questionnaires | To be assessed 5 months after start of study
Experiences of CHW about themselves as treatment providers assessed by indepth interviews using questionnaires | To be assessed 8 months after start of study
Perceptions and experiences of caregivers belonging to disadvantaged section of the community who could not access treatment from CHWs assessed by using questionnaires, indepth interviews | To be assessed at baseline
Perceptions and experiences of caregivers belonging to disadvantaged section of the community who could not access treatment from CHWs assessed by using questionnaires, indepth interviews | To be assessed 5 months after start of study
Perceptions and experiences of caregivers belonging to disadvantaged section of the community who could not access treatment from CHWs assessed by using questionnaires, indepth interviews | To be assessed 8 months after start of study
Proportion of caregivers who complied with referral. | To be assessed at baseline
Proportion of caregivers who complied with referral. | To be assessed 5 months after start of study
Proportion of caregivers who complied with referral. | To be assessed 8 months after start of study
Proportion of children treated by ANMs with injectable antibiotics. | To be assessed at baseline
Proportion of children treated by ANMs with injectable antibiotics. | To be assessed 5 months after start of study
Proportion of children treated by ANMs with injectable antibiotics. | To be assessed 8 months after start of study
Proportion of times of families who tried to contact CHW and were unable to do so. | To be assessed at baseline
Proportion of times of families who tried to contact CHW and were unable to do so. | To be assessed 5 months after start of study
Proportion of times of families who tried to contact CHW and were unable to do so. | To be assessed 8 months after start of study

CONTACTS AND LOCATIONS:
Overall Officials: Sarmila Mazumder, MBBS, PhD, Principal Investigator — Centre for Health Research and Development, Society for Applied Studies
Locations (1):
- CHRD, Society for Applied Studies, Palwal, Haryana, India